CLINICAL TRIAL: NCT00790595
Title: Phase I, Open Label, Single Center, Multiple Dose, Dose Escalation Clinical Study of SU011248 in Subjects With High Risk Prostate Cancer Who Have Elected to Undergo Radical Prostatectomy
Brief Title: Clinical Study of SU011248 in Subjects With High Risk Prostate Cancer Who Have Elected to Undergo Radical Prostatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-03-129; Pfizer2005-0958
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental): 5 Subjects will receive 37.5 mg/d of the study drug for 1 week.
  Interventions: Drug: SU011248
- Group B (Experimental): 5 Subjects will receive 50.0 mg/d of the study drug for 1 week.
  Interventions: Drug: SU011248
- Group C (Experimental): 5 Subjects will receive 37.5 mg/d of the study drug for 2 weeks.
  Interventions: Drug: SU011248
- Group D (Experimental): 5 Subjects will receive 50.0 mg/d of the study drug for 2 weeks.
  Interventions: Drug: SU011248
- Group E (Experimental): 5 Subjects will receive 50.0 mg/d of the study drug for 4 weeks.
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: SU011248 — 5 Subjects will receive 50.0 mg/d of the study drug for 2 weeks.
  Arms: Group D
Drug: SU011248 — 5 Subjects will receive 50.0 mg/d of the study drug for 4 weeks.
  Arms: Group E
Drug: SU011248 — 5 Subjects will receive 50.0 mg/d of the study drug for 1 week.
  Arms: Group B
Drug: SU011248 — 5 Subjects will receive 37.5 mg/d of the study drug for 1 week.
  Arms: Group A
Drug: SU011248 — 5 Subjects will receive 37.5 mg/d of the study drug for 2 weeks.
  Arms: Group C

SUMMARY:
Prostate cancer is prevalent in the United States, with approximately 230,110 new cases and 29,900 deaths in 2004. Approximately 30% of new cases will be clinical stage T3 when they are diagnosed. This is a stage in which there is high probability that the cancer has spread beyond the prostate gland itself, making it much more difficult to treat. In these cases, when surgery is done by itself and the prostate is removed, it is still very likely that some cancer that has spread beyond the prostate remains and will get worse. Radiation applied to the prostate also does not work well on tumors that have spread beyond the prostate. Even surgery and radiation combined have not eliminated the problems caused by prostate cancer that has spread into the tissue outside the prostate itself.

New treatments are needed to deal with prostate cancer at this more serious stage. Study doctors believe that it might be possible to shrink the prostate cancer using a new drug called SUO11248 or Sunitinib. After the patients take the drug, study doctors believe the cancer will shrink back to within the prostate, and they can then surgically remove the prostate and all the cancer. Patients on this study also will be given increasing doses of Sunitinib to find out how much of the drug can be given safely.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate glad.
* Informed of, willing, and able to comply with, the requirements of the investigational study and have signed a written informed consent in accordance with institutional regulatory guidelines.
* Subjects defined as being at high risk for disease relapse based on the following criteria: PSA > 10 ng/ml, and any one of the following: Gleason > 7 or T stage > T2b.
* Patients must have elected to and are a candidate to undergo a radical prostatectomy.
* Males greater than 18 years of age and less than or equal to 75 years of age (physiologic) any racial/ethnic group.
* Free of significant abnormal findings as determined by screening history, physical exam, vital signs (blood pressure, heart rate, respiration rate, and temperature), and urinalysis.
* Performance status: ECOG < 2.
* Life expectancy of at least 5 years.
* Absolute granulocyte count > 1,500/mm3.
* Platelet count > 100,000.
* Hemoglobin > 9.0 g/dL.
* Serum calcium < 12.0 mg/dL Adequate hepatic function as evidenced by ALT and AST values within normal range. Adequate organ function as defined by the following criteria: Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) < 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT < 5 x ULN if liver function abnormalities are due to underlying malignancy.
* Creatinine < 1.5 ULN.

Exclusion Criteria:

* Patients who have stage T2a or less prostate cancer, Gleason < 6, PSA <10-ng/mL.
* Prior hormonal, surgical, radiopharmaceutical or radiation therapy, cryotherapy, biological response modifiers, or systematic chemotherapy to treat prostatic carcinoma.
* Surgery within four weeks of study entry.
* Evidence of regional and/or distant metastases.
* Use of an investigational drug within 30 days prior to study entry.
* NCI CTCAE Version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment.
* Any of the following thing the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade > 2.
* Prolonged QTc interval on baseline EKG.
* Uncontrolled Hypertension (>150/100 mm Hg despite optimal medical therapy).
* Patients receiving CYP3A4 inducers or inhibitors; patients should not take grapefruit juice or St. John's Wort while on the study
* Known active infection.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of SU011248 by histological examination of prostate tumors following radical prostatectomy. | 24 months
To determine maximum tolerable dose of SU011248 when administered with prostate cancer prior to radical prostatectomy. | 4 weeks

SECONDARY OUTCOMES:
To evaluate the effects of SUO11248 on tumoral phospho VEGF/PDGF, receptor TK pathways, microvessel density, antiangiogenic activities and serum PSA levels. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Background] Weir HK, Thun MJ, Hankey BF, Ries LA, Howe HL, Wingo PA, Jemal A, Ward E, Anderson RN, Edwards BK. Annual report to the nation on the status of cancer, 1975-2000, featuring the uses of surveillance data for cancer prevention and control. J Natl Cancer Inst. 2003 Sep 3;95(17):1276-99. doi: 10.1093/jnci/djg040. PMID 12953083
- [Background] Cancer Facts and Figures 2004. American Cancer Society, 2004.
- [Background] Pound CR, Partin AW, Eisenberger MA, Chan DW, Pearson JD, Walsh PC. Natural history of progression after PSA elevation following radical prostatectomy. JAMA. 1999 May 5;281(17):1591-7. doi: 10.1001/jama.281.17.1591. PMID 10235151
- [Background] Roehl KA, Han M, Ramos CG, Antenor JA, Catalona WJ. Cancer progression and survival rates following anatomical radical retropubic prostatectomy in 3,478 consecutive patients: long-term results. J Urol. 2004 Sep;172(3):910-4. doi: 10.1097/01.ju.0000134888.22332.bb. PMID 15310996
- [Background] Kasamon KM, Dawson NA. Update on hormone-refractory prostate cancer. Curr Opin Urol. 2004 May;14(3):185-93. doi: 10.1097/00042307-200405000-00008. PMID 15069310
- [Background] Zagars GK. Prostate-specific antigen as a prognostic factor for prostate cancer treated by external beam radiotherapy. Int J Radiat Oncol Biol Phys. 1992;23(1):47-53. doi: 10.1016/0360-3016(92)90542-p. PMID 1374065
- [Background] Stamey TA, Kabalin JN, Ferrari M. Prostate specific antigen in the diagnosis and treatment of adenocarcinoma of the prostate. III. Radiation treated patients. J Urol. 1989 May;141(5):1084-7. doi: 10.1016/s0022-5347(17)41176-1. PMID 2468796
- [Background] Kabalin JN, Hodge KK, McNeal JE, Freiha FS, Stamey TA. Identification of residual cancer in the prostate following radiation therapy: role of transrectal ultrasound guided biopsy and prostate specific antigen. J Urol. 1989 Aug;142(2 Pt 1):326-31. doi: 10.1016/s0022-5347(17)38746-3. PMID 2473221
- [Background] Zagars GK, von Eschenbach AC, Johnson DE, Oswald MJ. Stage C adenocarcinoma of the prostate. An analysis of 551 patients treated with external beam radiation. Cancer. 1987 Oct 1;60(7):1489-99. doi: 10.1002/1097-0142(19871001)60:73.0.co;2-9. PMID 3113715
- [Background] Bagshaw MA, Cox RS, Ramback JE. Radiation therapy for localized prostate cancer. Justification by long-term follow-up. Urol Clin North Am. 1990 Nov;17(4):787-802. PMID 2219577
- [Background] Wheeler JA, Zagars GK, Ayala AG. Dedifferentiation of locally recurrent prostate cancer after radiation therapy. Evidence for tumor progression. Cancer. 1993 Jun 1;71(11):3783-7. doi: 10.1002/1097-0142(19930601)71:113.0.co;2-x. PMID 8490929
- [Background] Cumming JA, Ritchie AW, Goodman CM, McIntyre MA, Chisholm GD. De-differentiation with time in prostate cancer and the influence of treatment on the course of the disease. Br J Urol. 1990 Mar;65(3):271-4. doi: 10.1111/j.1464-410x.1990.tb14725.x. PMID 2337747
- [Background] Stamey TA and McNeal JE: Adenocarcinoma of the prostate. In Campbell's Urology 6th edition (Walsh PC, Retik AB, Stamey MA and Vaughan ED, eds), W.B. Saunders Co., pp 1159-1221, 1992.
- [Background] Stamey TA, Villers AA, McNeal JE, Link PC, Freiha FS. Positive surgical margins at radical prostatectomy: importance of the apical dissection. J Urol. 1990 Jun;143(6):1166-72; discussion 1172-3. doi: 10.1016/s0022-5347(17)40216-3. PMID 2342177
- [Background] Rosen MA, Goldstone L, Lapin S, Wheeler T, Scardino PT. Frequency and location of extracapsular extension and positive surgical margins in radical prostatectomy specimens. J Urol. 1992 Aug;148(2 Pt 1):331-7. doi: 10.1016/s0022-5347(17)36587-4. PMID 1635129
- [Background] Catalona WJ, Bigg SW. Nerve-sparing radical prostatectomy: evaluation of results after 250 patients. J Urol. 1990 Mar;143(3):538-43; discussion 544. doi: 10.1016/s0022-5347(17)40013-9. PMID 2304166
- [Background] Stein A, deKernion JB, Dorey F. Prostatic specific antigen related to clinical status 1 to 14 years after radical retropubic prostatectomy. Br J Urol. 1991 Jun;67(6):626-31. doi: 10.1111/j.1464-410x.1991.tb15228.x. PMID 1712655
- [Background] Frazier HA, Robertson JE, Humphrey PA, Paulson DF. Is prostate specific antigen of clinical importance in evaluating outcome after radical prostatectomy. J Urol. 1993 Mar;149(3):516-8. doi: 10.1016/s0022-5347(17)36132-3. PMID 7679755
- [Background] R Motzer, B Rini, M Michaelson, B Redman, G Hudes, G Wilding, R Bukowski, D George, S Kim, I Chen, C Baum and the SU11248 Study Group: Phase 2 Trials of SU11248 Show Antitumor Activity in Second-Line Therapy for Patients with Metastatic Renal Cell Carcinoma (RCC). ASCO, 2005.